CLINICAL TRIAL: NCT03368755
Title: Effect of Intrauterine Growth Restriction on Respiratory Muscle Function and Exercise Tolerance in Childhood
Brief Title: IUGR, Respiratory Muscle Function, and Exercise Capacity in Childhood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Patras (Other)
Collaborators: European Society for Paediatric Research (ESPR) (Unknown)
Responsible Party: Principal Investigator, Fouzas Sotirios, Pediatric Pulmonologist, Assistant Professor in Pediatrics, University of Patras
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IUGR-CPET_PATRAS
Record Dates: First submitted 2017-11-24; First posted 2017-12-11 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Intrauterine Growth Restriction; Cardiopulmonary Disease
MeSH Terms: conditions — Fetal Growth Retardation; Pulmonary Heart Disease | interventions — Exercise Test

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cases (IUGR) (Experimental): 50 school-aged children (7-10 years old) exposed to IUGR (birth weight <10th percentile & fetal ultrasound documentation) and of comparable gestational age with controls Intervention: Cardiopulmonary Exercise Testing and Respiratory Muscle Strength and Endurance
  Interventions: Diagnostic Test: Cardiopulmonary Exercise Testing; Diagnostic Test: Respiratory Muscle Strength and Endurance
- Controls (Active Comparator): 100 school-aged children (7-10 years old) not exposed to IUGR (birth weight <10th percentile & fetal ultrasound documentation) and of comparable gestational age with cases.
  Intervention: Cardiopulmonary Exercise Testing and Respiratory Muscle Strength and Endurance
  Interventions: Diagnostic Test: Cardiopulmonary Exercise Testing; Diagnostic Test: Respiratory Muscle Strength and Endurance

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary Exercise Testing — Pimax, Pemax, airway pressure at 100 msec after occlusion (P0.1), and Ti and Ttot will be measured by the Micro 5000 device (Medisoft, Sorinnes, Belgium). TTImus will be calculated as (Pimean / Pimax) x (Ti / Ttot), where Pimean is the mean airway pressure resulting from the formula Pimean = 5 x P0.1 x Ti9. RM function will be determined a) prior to CPET, b) during CPET when the anaerobic threshold (AT) will be reached, and c) after CPET, when heart rate (HR) and oxygen consumption will be normalized.
Diagnostic Test: Respiratory Muscle Strength and Endurance — CPET will be performed by the Ultima CPX system (Medgraphics, St. Paul, USA), using a cycle ergometer and according to a standardized protocol. The following parameters will be recorded: total work in Watts, maximum HR, maximum oxygen consumption (VO2max), AT indices (work, HR, VO2 ) and duration of recovery.

SUMMARY:
The study hypothesis is that intrauterine growth restriction (IUGR) may have long-term effects on respiratory muscle (RM) function, thus leading to reduced exercise capacity later in life. The objective is to investigate the above hypothesis by comparing RM function and cardiopulmonary exercise testing (CPET) parameters between school-aged children exposed to IUGR and healthy controls.

DETAILED DESCRIPTION:
Introduction

Epidemiological evidence supports the existence of a link between intrauterine growth restriction (IUGR) and reduced exercise capacity in young adulthood. Prolonged intrauterine hypoxia results in redistribution of fetal cardiac output towards the vital organs at the expense of skeletal muscles, and experimental data show that the muscles of animals exposed to IUGR may suffer permanent structural and functional changes. Prematurity, which often accompanies IUGR, is also associated with reduced exercise capacity later in life, supposedly due to airflow limitation, air trapping and/or reduced gas-exchange capacity.

The respiratory muscles (RM) play a central role in the development (and perception) of locomotor muscle fatigue, which represents the major determinant of exercise limitation in otherwise healthy subjects. Heavy and/or sustained respiratory work leads to accumulation of metabolites in RM and triggers reflexes that increase the sympathetic vasoconstrictor outflow to the skeletal muscles, thus promoting fatigue. In support of the above concept, targeted RM training has been shown to increase the fatigability threshold and improve exercise performance.

RM function can be assessed by means of strength and endurance, which can be estimated non-invasively by the maximum inspiratory and expiratory pressure (Pimax and Pemax), and the tension-time index (TTImus), respectively. TTImus is a composite parameter that reflects the balance between the capacity of RM and the load imposed upon them; high TTImus values indicate low endurance and increased risk of respiratory fatigue. In adults, impaired exercise tolerance is associated with reduced RM strength and endurance, both in normal and pathological conditions. However, similar data are not available in children.

Hypothesis and objectives

The study hypothesis is that IUGR may have long-term effects on RM function, thus leading to reduced exercise capacity later in life. Other factors, such as the presence and degree of respiratory dysfunction, the performance of the skeletal muscles and the nutritional status, may also be involved. The study objective is to investigate the above hypothesis by comparing RM function and cardiopulmonary exercise testing (CPET) parameters between school-aged children exposed to IUGR and healthy controls, taking also into account the aforementioned confounders.

Methods

Population

In this case-control study, 50 school-aged children (7-10 years old) exposed to IUGR (birth weight <10th percentile & fetal ultrasound documentation) will be compared with 100 matched for age and gestational age controls. The study will be performed in the Pediatric CPET laboratory of the University Hospital of Patras, Greece, during a 2-year period (2018-2020). Participants will be recruited from the long-term follow-up program offered to all children who are born preterm or with IUGR, and from the local schools (healthy full-term controls). The protocol will be approved by the hospital Ethics Committee and parental informed consent will be obtained prior to enrollment.

Protocol

After a thorough review of the medical history, participants will undergo the following tests:

1. Nutritional status, body composition and skeletal muscle strength. Initially, weight and height will be measured, and the body mass index (BMI) will be calculated. Body composition (muscular mass, body fat, water) will be determined by the InBody 270 Body Composition Analyzer (Biospace, Seoul, Korea) using bioelectrical impedance analysis. Skeletal muscle strength (grasping power) will be measured using a digital grip dynamometer (Grip-D, TAKEI, Japan).
2. Lung function measurements. Spirometry, measurement of lung volumes (helium dilution technique) and measurement of lung diffusion capacity for carbon monoxide (DLCO) will be performed prior to CPET using the Jaeger MasterScreen PFT device (CareFusion, San Diego, USA). Spirometric measurements will be repeated at 5, 10, and 15 minutes after CPET.
3. RM function. Pimax, Pemax, airway pressure at 100 msec after occlusion (P0.1), and Ti and Ttot will be measured by the Micro 5000 device (Medisoft, Sorinnes, Belgium) according to the guidelines. TTImus will be calculated as (Pimean / Pimax) x (Ti / Ttot), where Pimean is the mean airway pressure resulting from the formula Pimean = 5 x P0.1 x Ti. RM function will be determined a) prior to CPET, b) during CPET when the anaerobic threshold (AT) will be reached, and c) after CPET, when heart rate (HR) and oxygen consumption will be normalized (recovery period).
4. CPET. CPET will be performed by the Ultima CPX system (Medgraphics, St. Paul, USA), using a cycle ergometer and according to a standardized protocol11 and the established guidelines. The following parameters will be recorded: total work in Watts, maximum HR, maximum oxygen consumption (VO2max), AT indices (work, HR, VO2 ) and duration of recovery.

Statistical analysis

Between-group comparisons will be performed with Student's t or Mann-Whitney U test, as appropriate. Linear regression analysis will be used to explore the relationship between RM function and CPET parameters, after adjustment for nutritional status, body composition, lung function, and prematurity. The trend of Pimax, Pemax, and TTImus changes during CPET (baseline - AT - recovery) will be also assessed and compared between groups. The analyses will be performed using the IBM SPSS version 23.0 (IBM Corp., Armonk, NY).

Innovation and implications

The study will be the first to explore whether IUGR is associated with impaired exercise tolerance in childhood due to RM dysfunction, while taking into account the confounding effect of prematurity, impaired lung function, body composition and nutritional status.

Should the relationship IUGR - RM dysfunction - exercise limitation be confirmed, it will provide new insights on the long-term effects of IUGR; impaired exercise tolerance may lead to reduced physical activity, thus enhancing the well-known metabolic and cardiovascular consequences of IUGR later in life. In this regard, the findings of this study may assist in identifying children at risk and planning targeted strategies to improve exercise capacity in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* (Cases) School-aged children (7-10 years old) exposed to IUGR (birth weight <10th percentile & fetal ultrasound documentation)
* (Controls) School-aged children (7-10 years old) NOT exposed to IUGR (birth weight >10th percentile)

Exclusion Criteria:

* Disability
* Congenital heart disease
* Current (active) respiratory infection

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
VO2 max | 1 day (during exercise testing)
  Maximum O2 consumption, in ml/kg/min. The index will be compared between IUGR and controls.
TTmus | 1 day (during exercise testing)
  Tension-time index of the respiratory muscles. No values (ratio). The index will be compared between IUGR and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Sotirios Fouzas, MD, PhD, Principal Investigator — University of Patras, Greece; Gabriel Dimitriou, MD, PhD, Study Chair — University of Patras, Greece
Locations (1):
- University Hospital of Patras, Pátrai, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Svedenkrans J, Henckel E, Kowalski J, Norman M, Bohlin K. Long-term impact of preterm birth on exercise capacity in healthy young men: a national population-based cohort study. PLoS One. 2013 Dec 6;8(12):e80869. doi: 10.1371/journal.pone.0080869. eCollection 2013. PMID 24324639
- [Background] Rosenberg A. The IUGR newborn. Semin Perinatol. 2008 Jun;32(3):219-24. doi: 10.1053/j.semperi.2007.11.003. PMID 18482625
- [Background] Lane RH, Chandorkar AK, Flozak AS, Simmons RA. Intrauterine growth retardation alters mitochondrial gene expression and function in fetal and juvenile rat skeletal muscle. Pediatr Res. 1998 May;43(5):563-70. doi: 10.1203/00006450-199805000-00001. PMID 9585000
- [Background] Lane RH, Maclennan NK, Daood MJ, Hsu JL, Janke SM, Pham TD, Puri AR, Watchko JF. IUGR alters postnatal rat skeletal muscle peroxisome proliferator-activated receptor-gamma coactivator-1 gene expression in a fiber specific manner. Pediatr Res. 2003 Jun;53(6):994-1000. doi: 10.1203/01.PDR.0000064583.40495.51. Epub 2003 Mar 19. PMID 12646730
- [Background] Kilbride HW, Gelatt MC, Sabath RJ. Pulmonary function and exercise capacity for ELBW survivors in preadolescence: effect of neonatal chronic lung disease. J Pediatr. 2003 Oct;143(4):488-93. doi: 10.1067/S0022-3476(03)00413-X. PMID 14571227
- [Background] Dempsey JA, Romer L, Rodman J, Miller J, Smith C. Consequences of exercise-induced respiratory muscle work. Respir Physiol Neurobiol. 2006 Apr 28;151(2-3):242-50. doi: 10.1016/j.resp.2005.12.015. PMID 16616716
- [Background] Regamey N, Moeller A. Paediatric exercise testing. Eur Respir Mon 2010; 47: 291-309
- [Background] McConnell AK. CrossTalk opposing view: respiratory muscle training does improve exercise tolerance. J Physiol. 2012 Aug 1;590(15):3397-8; discussion 3399-400. doi: 10.1113/jphysiol.2012.235572. No abstract available. PMID 22855045
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Foglio K, Clini E, Facchetti D, Vitacca M, Marangoni S, Bonomelli M, Ambrosino N. Respiratory muscle function and exercise capacity in multiple sclerosis. Eur Respir J. 1994 Jan;7(1):23-8. doi: 10.1183/09031936.94.07010023. PMID 8143827
- [Background] Godfrey S. Exercise Testing in Children. London, UK: WB Saunders Company Ltd., 1974.
- [Background] Ross MG, Beall MH. Adult sequelae of intrauterine growth restriction. Semin Perinatol. 2008 Jun;32(3):213-8. doi: 10.1053/j.semperi.2007.11.005. PMID 18482624